CLINICAL TRIAL: NCT01539980
Title: Clinical Efficacy of Wound Dressing Containing Silk Sericin for Split-thickness Skin Graft Donor Site Treatment
Brief Title: Clinical Study on Silk Sericin Wound Dressing for Split-thickness Skin Graft Donor Sites Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Associate Professor, Chulalongkorn University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NRCT-2554-21
Record Dates: First submitted 2012-02-17; First posted 2012-02-28 (Estimated); Results first posted 2015-04-02 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-04

CONDITIONS: Late Complication From Skin Graft; Infection of Skin Donor Site; Impaired Wound Healing; Pain, Intractable
Keywords: Sericin scaffold; Wound healing; Skin graft donor
MeSH Terms: conditions — Pain, Intractable

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sericin scaffold (Experimental)
  Interventions: Device: Sericin scaffold

INTERVENTIONS:
Device: Sericin scaffold — Device: wound dressing containing silk sericin A scaffold from silk sericin-polyvinyl alcohol-glycerin blending are applied on one half of the skin graft donor site Device: fine mesh gauze impregnated with paraffin and 0.5%chlorhexidine acetate (Bactigras, Smith&Nephew, London, UK) are applied on the other half of the skin graft donor site

SUMMARY:
1. Silk sericin wound dressing may reduce time for complete epithelialisation of split-thickness skin graft donor sites compared to Bactigras®.
2. Silk sericin wound dressing may reduce pain level at split-thickness skin graft donor sites compared to Bactigras® .
3. Silk sericin wound dressing may not cause split-thickness skin graft donor sites infection as compared to Bactigras®.
4. Split-thickness skin graft donor sites which treat by silk sericin wound dressing may not cause significant adverse events.

DETAILED DESCRIPTION:
Split-thickness skin graft (STSG) is a surgical procedure to repair losses of skin by transferring of a section of healthy skin (donor site) to replace the damaged tissue in another area of the body (recipient site). However, the patients will have a new wound at donor sites which need appropriate wound dressing to increase healing and reduce complications. Since silk sericin can form a dressing which can accelerate wound healing process and protect wound from environment, the aim of this study is to investigate how well silk sericin wound dressing cures STSG donor sites by comparing to Bactigras® which is a commonly used paraffin-impregnated fine mesh gauze. Silk sericin wound dressing is a promising material which can shorten the treatment course and reduce pain for the patients who have donor sites. This study design is a single-center, randomized, open and paralleled positive control study.18-60- year-old patients of both genders who undergo STSG at anterolateral thigh in Division of plastic and reconstructive surgery, King Chulalongkorn Memorial Hospital from April 2012 to January 2013 will be recruited in the study. The thickness of donor sites fall between 0.15-0.45 mm (0.006-0.018 inches) and their sizes are at least 100 cm2. The exclusion criteria are donor sites other than thigh or located at high risk of infection. Patients who are immunocompromised or mental defect, who are unlikely to comply with protocol or pregnant or lactating or known hypersensitivity to the investigational products are also excluded. All subjects sign the informed consents after an overall discussion of the protocol, its rationale and the potential risks. Donor sites are equally divided into 2 parts; upper and lower part of the leg. Using a random number table allocation, silk sericin wound dressing is randomly applied on one half and the other half will be covered by Bactigras®. Postoperatively, surgeons will observe all donor sites daily for treatment evaluation and any possible local adverse events without removing the primary dressings, except there is excessive fluid leakage or any sign of infection. Patients assess for pain level in every observations by using Visual Analog Scale. Time for complete epithelialisation is duration between finishing surgical procedure and the dressing spontaneously peeling off from donor sites without causing pain. If there is any sign of infection such as swelling, edema, purulent discharge, bad odor, a swab evaluation at the suspected area will be done to find an appropriate management. Blood sample will be collected from patients pre- and postoperatively (with in 24h, day3 and before patient discharge) for CBC, blood glucose, electrolyte, hepatic and renal function analysis and proinflammatory cytokine measurement. This study may show any possible adverse events, both local and systemic effect, caused by silk sericin dressing. Proinflammatory cytokines patterns of the patients underwent STSG will be revealed in this study which may be relate to clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-60 years
* Patients who require STSG such as burn, trauma, venous ulcers, or surgical removal of cutaneous malignancies etc.
* Patients whom surgeons assess that ready for undergoing STSG
* Sufficient normal skin at anterolateral thigh area for 1 or more STSG donor sites
* The thickness of donor sites fall between 0.15-0.45 mm (0.006-0.018 inches) and their sizes are at least 100 cm2
* Patients who are willing to participate in the trial and to sign the informed consent form.

Exclusion Criteria:

* Use others area for STSG donor sites other than thigh
* Donor sites are located at high risk of infection such as harvesting closed to current infective wound (excessive purulent discharge or bad odor)
* Patients who are immunocompromised or mental defect
* Patients who cannot or not willing to comply with the study protocol
* Known allergy or hypersensitivity reaction to silk sericin or chlorhexidine acetate
* Pregnancy or lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-08; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chulalongkorn Hospital, Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sericin Scaffold
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sericin Scaffold
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 12
Region of Enrollment [Number; unit: participants]
  Thailand | 30
Wound size [Mean (Standard Deviation); unit: square centrimeter] | 124.74 (86.72)
Body temperature [Mean (Standard Deviation); unit: Degree celcius] | 36.73 (0.37)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Efficacy of Wound Dressing Containing Silk Sericin for Split-thickness Skin Graft Donor Site Treatment
Description: Time for complete epithalization is duration between finishing surgical procedure and the dressing spontaneously peeling off from donor sites without causing pain. The wounds completely close and without fluid leakage and are able to exposed to the environment without pain. This duration should not exceed than 14 days.
Time Frame: Within 14 days after operation
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Sericin Scaffold
Number analyzed (Participants) | 30
Days | 12 (5)

2. Secondary Outcome: Clinical Safety of Wound Dressing Containing Silk Sericin for Split-thickness Skin Graft Donor Site Treatment
Description: Number of patients with infected wound
Time Frame: Within 14 days after operation
Measure: Number; unit: Number of patients with infected wound
Arm/Group | Sericin Scaffold
Number analyzed (Participants) | 30
Number of patients with infected wound | 0

3. Secondary Outcome: Pain Levels of Wounds
Description: Pain may occur on operation wounds. Visual analog scale is used by patients themselves for monitoring the pain level with 0 = no pain, 10 = worst possible pain.
Time Frame: Within 14 days after operation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sericin Scaffold
Number analyzed (Participants) | 30
units on a scale | 2.60 (1.40)

4. Secondary Outcome: Proinflammatory Cytokines (IL)
Description: The proinflammatory cytokines from wound exudate will be measured for predicting the inflammatory level. ELISA kit is used.
Time Frame: Within 14 days after operation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sericin Scaffold
Number analyzed (Participants) | 30
pg/mL | 31.65 (16.71)

5. Secondary Outcome: Liver Enzyme (AST)
Description: Large, open wound may absorb some materials from wound dressing. If those materials are toxic, liver enzyme (a major organ for elimination of any toxicities) will be increased.
Time Frame: Within 14 days after operation
Measure: Mean (Standard Deviation); unit: u/L
Arm/Group | Sericin Scaffold
Number analyzed (Participants) | 30
u/L | 19 (10)

ADVERSE EVENTS:
Arm/Group | Sericin Scaffold
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 2/30
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sericin Scaffold (N=30)
Itching (Skin and subcutaneous tissue disorders) | 2 (2) — Patients may experience itching around the operation wounds

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No